CLINICAL TRIAL: NCT00206466
Title: A Randomized Multicenter Trial of Neoadjuvant Taxotere and Adriamycin/Cytoxan(AC): A Biologic Correlative Study
Brief Title: Biologic Correlative Taxotere/AC
Acronym: TAX/AC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Breast Care Center (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-11624
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: neoadjuvant; chemosensitivity; chemotherapy; breast cancer; tumor; taxotere; AC
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Docetaxel; Doxorubicin; Cyclophosphamide

ARMS (1):
- One (Active Comparator): Taxotere
  Interventions: Drug: Taxotere; Drug: Adriamycin/cytoxan

INTERVENTIONS:
Drug: Taxotere — Docetaxel (Taxotere) 100 mg/m2 is to be administered on day 1. A core biopsy is to be performed one day after chemotherapy (day 2) and on days 8, 15 and 22. On day 22, after repeat core biopsy, a second cycle of docetaxel (Taxotere) chemotherapy (100 mg/m2) will be given. Docetaxel (Taxotere) will be given three-weekly for a total of four cycles. Primary surgery will then be conducted, if operable, following completion of neoadjuvant treatment. Adjuvant AC (doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2, every three weeks) for four cycles will then be administered. Adjuvant radiotherapy will be considered following completion of AC chemotherapy. Patients whose tumors were ER and/or PgR positive would be commenced on tamoxifen for five years after completion of AC chemotherapy.
  Other Names: Docetaxel (Taxotere)
Drug: Adriamycin/cytoxan — Adjuvant AC (doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2, every three weeks) for four cycles will then be administered. Adjuvant radiotherapy will be considered following completion of AC chemotherapy. Patients whose tumors were ER and/or PgR positive would be commenced on tamoxifen for five years after completion of AC chemotherapy.
  Other Names: doxorubicin 60 mg/m2 and cyclosphosphamide 600 mg/m2

SUMMARY:
We are asking you to take part in a research study of biomarkers (characteristics or traits of the genes inside cancer cells). We want to learn if these biomarkers could help us learn how well your breast cancer may respond (improve) to chemotherapy (drugs to treat cancer).

DETAILED DESCRIPTION:
Breast cancer and systemic chemotherapy: Systemic chemotherapy for operable breast cancer significantly decreases the risk of relapse and death. However, it is not possible to identify those patients at the outset who are likely to respond to adjuvant treatment and which type of treatment should be used. Adjuvant treatment given before surgery (neoadjuvant therapy) has a number of advantages in breast cancer, including a reduction in the requirement for mastectomy. Access to the primary tumor during early treatment allows for in vivo testing for predictive markers obtained by core biopsies that occur with successful treatment.

Predictive markers in breast cancer: Prognostic factors like tumor size and nodal involvement are important indicators for breast cancer survival but have not been shown to be predictive of sensitivity to chemotherapy. With endocrine therapy, the prime example of a predictive marker is estrogen receptor (ER) expression, which predicts for response to tamoxifen and other endocrine treatments. However, predictive markers for chemotherapy are not established. Overexpression of c-erbB-2 might be associated with decreased response to CMF and increased response to anthracycline-based treatment, but these observations are still contentious. Expression of topoisomerase II may also reflect responsiveness to anthracycline chemotherapy. Recently, some emerging data also suggest that c-erbB2 may be a marker of taxane sensitivity. As such, we lack predictive biomarkers that could give early information on how effective chemotherapy is and whether additional treatment might be beneficial. A test for chemotherapy sensitivity, equivalent to ER in predicting response to endocrine therapy, would greatly facilitate treatment decisions so that in an ideal scenario, the treatment of each individual patient could be based on specific features of her disease.

Neoadjuvant chemotherapy: Preoperative chemotherapy for large tumors (>3cm) or inoperable breast cancer is well established and is the standard of care for locally advanced breast cancer. Data from large series of patients have demonstrated that preoperative (neoadjuvant) chemotherapy leads to significant reduction of tumor size (downstaging) and improves both the rate and the cosmetic results of breast-conserving surgery. A recent large randomized trial involving 1,523 patients compared preoperative and postoperative chemotherapy (NSABP B-18). Although results of this study have shown no difference in disease-free survival and survival in women on preoperative or postoperative doxorubicin and cyclophosphamide chemotherapy, significant downstaging of tumors was achieved so that more patients who received preoperative therapy were able to undergo breast-conserving surgery. The rate of breast conservation in NSABP B-18 was 85% in patients with tumors greater than 3 cm, with less than 5% of patients reported to have progressive disease while receiving neoadjuvant chemotherapy.

cDNA arrays: High-Throughput Quantitative Profiling of Gene Expression: With the advent of high-throughput quantitation of gene expression and cDNA technology, it is now possible to study expression of many genes simultaneously to characterize expression patterns in different breast cancers that may distinguish molecular phenotypes associated with clinical response to a treatment. In a recent report, a molecular classification of leukemia was demonstrated. Bone marrow aspirates taken from 38 patients with acute leukemia were evaluated for expression of 6,817 human genes. The 50 best discriminating genes were used to create a predictive index that was then applied to new samples and was found to accurately assign them as AML or ALL.

Preliminary data for differential patterns of gene expression in responders vs non-responders of Taxotere chemotherapy: We conducted a pilot study to investigate gene expression patterns on core biopsies of human breast cancers in responders and non-responders to Taxotere chemotherapy.

RNA was isolated from core biopsies of primary breast cancers taken from women before initiation of Taxotere chemotherapy. Clinical response was assessed after 12 weeks of treatment. We compared patterns of gene expression statistically in order to identify genes differentially expressed between responders and non-responders to this single chemotherapeutic agent.

Overall, these genes efficiently cluster tumors into 3 groups: CR, PR, and NR. We have selected 2337 genes from these data for further analysis. As expected, the majority of these genes show heterogeneous expression patterns independent of treatment response, but six large gene clusters (approximately 180 genes) appear to predict likelihood of response to Taxotere therapy. Consistent with an apoptosis-induction mode of action for taxanes, responsive tumors appear to have higher expression of stress-related proteins, such as mitochondrial proteins involved in apoptosis (cytochromes, proteasome subunits), and higher levels of motility-related microfilament proteins (actin, myosin, and tropomyosin). Non-responders patterns are more complex but show elevated levels of some microtubule proteins presumed to be targets of Taxotere therapy (tubulins, tubulin-interacting proteins) and elevated levels of inflammatory-response genes. Surprisingly, non-responders also showed elevated proliferation (KI67) and oncogene (ABL1, MYC and JUNB) expression levels. This molecular portrait of Taxotere resistance differs from the expected profiles of general chemoresistance. Quantitative RT-PCR and immunohistochemistry studies to confirm these differential gene patterns of expression are in progress for all 40 patients.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be female.
2. Signed informed consent.
3. Primary breast cancers must be of clinical and/or radiologic size >3 cm, and deemed surgically operable.
4. Negative serum pregnancy test (bHCG) within 7 days of starting study, if of child-bearing potential.
5. Adequate bone marrow function: Hematocrit of greater than 30%, total neutrophil count must be >1.5 x 109/L and platelets of > 100 x 109/L prior to the start of any cycle.
6. Renal function tests: creatinine within 1.5 times of the institution's upper limit of normal (ULN).
7. Liver function tests: Total serum bilirubin within ULN, and liver transaminases within 2.5 times ULN, and alkaline phosphatase within 5 times ULN.
8. Electrocardiogram showing no acute ischemic changes.
9. Performance status (WHO scale) <2.
10. Age > 18 years.
11. Patients older than 70 years of age should have left ventricular ejection fraction within ULN by MUGA or 2D Echocardiogram.

Exclusion Criteria:

1. Patients with metastatic breast cancer.
2. Pregnancy or unwillingness to use a reliable contraceptive method in women of child-bearing potential.
3. Women who are lactating or breastfeeding.
4. Severe underlying chronic illness or disease.
5. Peripheral neuropathy - grade 2 or greater.
6. Patients on other investigational drugs while on study will be excluded.
7. Severe or uncontrolled hypertension, history of congestive heart failure, acute myocardial infarction, or severe coronary arterial disease.
8. Prior taxane or anthracycline chemotherapy for malignancy.
9. Patients with a history of severe hypersensitivity reaction to Taxotere or other drugs formulated with polysorbate 80.
10. No previous or current malignancies at other sites within the last 5 years, with exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-04; Primary Completion 2006-04 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The primary objective this extension study is to obtain enough additional cases evaluable for microarray analyses to complete our studies to identify profiles of a small number of genes that are predictive of response. | 10 years

SECONDARY OUTCOMES:
To determine pathologic complete response and to correlate this to a prospectively determined Taxotere gene expression profile;time to tumor progression;overall survival | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar C Rimawi, MD, Principal Investigator — Baylor Breast Center
Locations (1):
- Baylor Breast Center, Houston, Texas, United States

REFERENCES:
- See also: Web Site — http://www.breastcenter.tmc.edu